CLINICAL TRIAL: NCT02981940
Title: A Phase 0/2 Study of Abemaciclib in Recurrent Glioblastoma
Brief Title: A Study of Abemaciclib in Recurrent Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Eudocia Quant Lee, MD, MD, MPH, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16-383
Record Dates: First submitted 2016-10-07; First posted 2016-12-05 (Estimated); Results first posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma
Keywords: Brain Tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — abemaciclib; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Abemaciclib with Surgery (Experimental): * Abemaciclib will be administered on a continuous twice daily dosing schedule
  * Patients who require re-operation will receive a short preoperative course of Abemaciclib
  * Tissue will be used to investigate the ability of Abemaciclib to pass through the blood brain barrier.
  * After recovery from surgery, participants will resume Abemaciclib. Each cycle lasts 28 days.
  * NOTE: enrollment to this arm is complete
  Interventions: Drug: Abemaciclib; Procedure: Surgery
- Abemaciclib without Surgery (Experimental): * Abemaciclib will be administered on a continuous twice daily dosing schedule. Each Cycle last 28 days.
  * NOTE: enrollment to this arm is complete
  Interventions: Drug: Abemaciclib
- Cohort 1 Surgery Arm (Experimental): Participants who require reoperation will be treated with abemaciclib for 10-14 days prior to surgery. Tissue will be used to further investigate the abilities of Abemaciclib. After surgery participants will come off study and pursue standard of care treatments at their treating physician's discretion.
  Interventions: Drug: Abemaciclib; Procedure: Surgery

INTERVENTIONS:
Drug: Abemaciclib — Abemaciclib capsule
  Other Names: LY2835219
Procedure: Surgery — Surgery
  Arms: Abemaciclib with Surgery; Cohort 1 Surgery Arm

SUMMARY:
This research study is studying a targeted therapy as a possible treatment for recurrent glioblastoma (GBM).

The following intervention will be used in this study:

-Abemaciclib

DETAILED DESCRIPTION:
This research study is a Phase 0/II clinical trial. Phase 0 clinical trials use only a few small doses of a drug. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved abemaciclib as a treatment for any disease.

Many brain cancers show over expression of a protein called cyclin D1. That means that the body makes too much cyclin D1, which affects enzymes called CDK 4 and CDK 6. Enzymes are substances in the body that help reactions between cells happen. Too much cyclin D1 triggers CDK 4 and CDK 6 to make more cells than normal. This extra cell production leads to the growth of tumors.

In laboratory studies, Abemaciclib was able to enter the brain, stop CDK 4 and CDK 6 from making cells, and slow growth of mice Glioblastoma.

In this research study, the investigators are looking to see how safe and effect Abemaciclib is with the participant type of cancer. In the surgical participants, the investigators are looking to see if Abemaciclib reached the brain tumor.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to understand and willing to sign a written informed consent document.
* Participants must be able to adhere to the dosing and visit schedules, and agree to record medication times accurately and consistently in a daily diary.
* Participants must be at least 18 years old on day of signing informed consent.
* Participants must have a Karnofsky Performance Status (KPS) ≥ 60
* Participants must be able to swallow capsules/tablets
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy of the trial are eligible.

Nature of illness and treatment history

* Participants must undergo central pathology review to histologically confirm the diagnosis of glioblastoma, IDH-wildtype; glioblastoma variants; or astrocytoma, IDH-mutant, WHO grade 4 (1 unstained slide or 1 H&E slide must be submitted to and reviewed by a pathologist at the DFCI Coordinating Center prior to enrollment of the participant for central pathology review).
* To be eligible for the study all participants (Cohort 1 and 2) are required to provide genomic profiling data from assays performed in a CLIA-certified lab. A sequencing-based assay is required and must include reporting of the RB1 gene in explicit terms within the report. Only sequencing assays that include coverage of all exons of the RB1 gene are able to be utilized (most commonly called a targeted exome assay; e.g. Oncopanel, Impact, FoundationOne). In addition, patients must provide a report of copy assessment which reports status of RB1. The reporting may be from a copy array (ideally Oncoscan SNP array or Agilent array CGH) or can also be from sequencing assay if copy status is explicitly provided with quantitative information regarding the status of relevant genes. Specifically, the reporting should provide the following information with respect to relevant biomarkers required for enrollment to the study as listed below.
* Results from genomic profiling must be sent to the DFCI Coordinating Center prior to enrollment of the participant for central pathology review.

  * Inactivation of CDKN2A/B or C in the tumor by homozygous deletion (evidence for more than single copy loss for any of the genes defined as array CGH/SNP log2 ratio of <0.3 by array CGH; or from sequencing data with sufficient coverage for evaluation). Rearrangement/evidence or intragenic breaks by copy or sequencing assay also will be considered eligible for study (any copy status).
  * OR
  * CDK4 or CDK6 high-level amplification. (The amplicon size must be <10Mb and the magnitude the gain must be log2 ratio >1.5 or estimated as >10 copies).
  * AND
  * Validation of wild-type RB status (no deletion/losses more than single copy by copy number or sequencing data; and/or no inactivating mutations by sequencing).
* Participants must be at first relapse of GBM. Relapse is defined as progression following initial therapy (i.e. radiation+/- chemo if that was used as initial therapy). The intent therefore is that patients had no more than 1 prior therapy (initial treatment). If the patient had a surgical resection for relapsed disease and no anti-cancer therapy was instituted for up to 12 weeks, and the patient undergoes another surgical resection, this is considered to constitute 1 relapse.
* Participants must have shown unequivocal evidence for tumor progression by MRI or CT scan.

  * For Cohort 2 subjects, CT or MRI within 14 days prior to study registration. For Cohort 2, corticosteroid dose must be stable or decreasing for at least 5 days prior to the scan. If steroids are added or the steroid dose is increased between the date of the screening MRI or CT scan and the start of treatment, a new baseline MRI or CT is required.
  * For Cohort 1 subjects, CT or MRI should be performed ideally within 14 days prior to study registration, but because the screening MRI for this subset of subjects will not be used for evaluation of response, it is acceptable for this MRI/CT to have been performed greater than 14 days prior to registration if unavoidable. Furthermore, for this same reason, fluctuation in corticosteroid dose around this MRI does not warrant repeat scan so long as there is documented unequivocal evidence of tumor progression available.
  * For Cohort 1 subjects, there must be > 2cm2 enhancing tissue available for resection and submission for study correlatives as determined by local treating team.
* Confirmation of availability of sufficient tissue from a prior surgery for correlative studies is required prior to enrollment; these samples must be sent to the DFCI Coordinating Center within 60 days of registration. Cohort 1 participants must have sufficient FFPE tissue from any surgery. Cohort 2 participants must have tissue from biopsy or resection from the most recent recurrence surgery.
* The following amount of archived tissue is required:

  * 20 unstained formalin fixed paraffin embedded (FFPE) sections (standard 4-5 micrometer thickness)
  * NOTE: if the above-mentioned tissue is not available from the most recent surgery revealing GBM, participants may be enrolled with tissue available from any prior surgery revealing GBM with prospective approval from the Overall PI.
* An interval of at least 12 weeks from the completion of radiation therapy to start of study drug unless there is a new area of enhancement consistent with recurrent tumor outside the radiation field (defined as the region outside the high-dose region or 80% isodose line) or there is unequivocal histologic confirmation of tumor progression.
* Participants must have recovered to grade 0 or 1 or pre-treatment baseline from clinically significant toxic effects of prior therapy (including but not limited to exceptions of alopecia, laboratory values listed per inclusion criteria, and lymphopenia which is common after therapy with temozolomide).
* From the projected start of scheduled study treatment, the following time periods must have elapsed:

  * 4 weeks or 5 half-lives (whichever is shorter) from any investigational agent;
  * 4 weeks from cytotoxic therapy (except 23 days for temozolomide; 6 weeks from nitrosoureas);
  * 4 weeks from antibodies;
  * 4 weeks or 5 half-lives (whichever is shorter) from other anti-tumor therapies.
  * 2 days from Novo-TTF
* Participants with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of progressive disease based upon nuclear imaging, MR spectroscopy, perfusion imaging or histopathology.
* Participants having undergone recent resection or open biopsy or stereotactic biopsy of recurrent or progressive tumor will be eligible for Cohort 2 as long as the following conditions apply:

  * They have recovered from the effects of surgery.
  * Residual disease following resection of recurrent tumor is not mandated for eligibility. To best assess the extent of residual disease post-operatively, an MRI or CT scan should ideally have been performed no later than 96 hours following surgery, or at least 28 days post-operatively, but scans performed outside of this window are considered acceptable if no alternative is available. In either case, the baseline/screening MRI must be performed within 14 days prior to registration. If the participant is taking corticosteroids, the dose must be stable or decreasing for at least 5 days prior to the scan. If steroids are added or the steroid dose is increased between the date of the screening MRI or CT scan and the start of treatment, a new baseline MRI or CT is required.

Clinical labs - performed within 14 days prior to registration

* Hematology:

  * Absolute neutrophil count (ANC) ≥ 1.5 x K/µL
  * Platelet count ≥ 100 x K/µL
  * Hemoglobin ≥ 8.0 g/dL
* Biochemistry:

  * Total serum calcium (corrected for serum albumin as needed) or ionized calcium within institution's normal range.
  * Magnesium within institution's normal range.
  * AST (SGOT) and ALT (SGPT) ≤ 3.0 x institution's ULN
  * Serum bilirubin ≤ 1.5 x institution's ULN
  * Serum creatinine ≤ 1.5 x institution's ULN or calculated 24-hour creatinine clearance ≥ 50 mL/min
  * Serum amylase ≤ 1.5 x institution's ULN
  * Serum lipase ≤ 1.5 x institution's ULN
* Coagulation studies:

  * INR < 2.0
  * PTT ≤ institution's ULN, unless receiving therapeutic low molecular weight heparin or oral factor Xa inhibitors Pregnancy and Reproduction
* The effects of abemaciclib on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) must agree to use a medically approved contraceptive method during the treatment period and for 3 months following the last dose of abemaciclib. Men must agree to use a reliable method of birth control and to not donate sperm during the study and for at least 3 months following the last dose of abemaciclib. Contraceptive methods may include an intrauterine device [IUD] or barrier method. If condoms are used as a barrier method, a spermicidal agent should be added as a double barrier protection.
* NOTE: Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Women of child-bearing potential must have a negative serum pregnancy test within 7 days prior to first dose of abemaciclib .

Exclusion Criteria:

Pathology

* Prior evidence of 1p/19q co-deletion.
* IDH1/2 mutation in any prior biopsy.

Previous therapies

* Participants who have received prior treatment with a CDK4/6 inhibitor.
* Participants who have received anti-VEGF targeted agents (e.g. bevacizumab, cediranib, aflibercept, vandetanib, XL184, sunitinib etc).

Concomitant medications

* Participants taking an enzyme-inducing anti-epileptic drug (EIAED): phenobarbital, phenytoin, fosphenytoin, primidone, carbamazepine, oxcarbazepine, eslicarbazepine, rufinamide, and felbamate. Participants must be off any EIAEDs for at least 14 days prior to starting study drug. A list of EIAEDs and other inducers of CYP3A4 can be found.
* Participants taking a drug known to be a strong inhibitor or inducer of isoenzyme CYP3A . Participant must be off CYP3A inhibitors and inducers for at least 14 days prior to starting study drug. NOTE: participants must avoid consumption of Seville oranges (and juice), grapefruits or grapefruit juice, grapefruit hybrids, pummelos and exotic citrus fruits from 7 days prior to the first dose of study drug and during the entire study treatment period due to potential CYP3A4 interaction.
* Participants receiving any other investigational agents.
* Current use of herbal preparations/medications, including but not limited to: St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, ginseng. Participants should stop using these herbal medications 7 days prior to first dose of study drug.
* Current use of warfarin sodium or any other coumadin-derivative anticoagulant. Participants must be off Coumadin-derivative anticoagulants for at least 7 days prior to starting study drug. Low molecular weight heparin is allowed.
* Requires treatment with high dose systemic corticosteroids defined as dexamethasone > 4 mg/day or bioequivalent for at least 3 consecutive days within 2 weeks of registration.

Other illnesses

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to abemaciclib.
* History of intratumoral or peritumoral hemorrhage if deemed significant by the treating investigator. If there are questions, the treating investigator should contact the study Overall P.I., Eudocia Quant Lee, MD, at 617-632-2166 or eqlee@partners.org.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, chronic liver disease (e.g., cirrhosis, hepatitis), chronic renal disease, pancreatitis, chronic pulmonary disease, or psychiatric illness/social situations that would limit compliance with study requirements. Subjects must be free of any clinically relevant disease (other than glioma) that would, in the treating investigator's opinion, interfere with the conduct of the study or study evaluations.
* Participant has an active systemic fungal and/or known viral infection (for example, human immunodeficiency virus antibodies, hepatitis B surface antigen or hepatitis C antibodies).
* Participants with diarrhea ≥ CTCAE grade 2
* Participant has active cardiac disease including any of the following:

  * Angina pectoris that requires the use of anti-anginal medications
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular and nodal arrythmias requiring a pacemaker or not controlled with medication
  * Conduction abnormality requiring a pacemaker
  * Valvular disease with document compromise in cardiac function
  * Symptomatic pericarditis
* Participant has a history of cardiac dysfunction including any of the following:

  * Myocardial infarction within the last 6 months prior to start of study drug, documents by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV, see Appendix B)
  * Documented cardiomyopathy
  * Congenital long QT syndrome
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of abemaciclib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or extensive small bowel resection). Participants with unresolved diarrhea ≥ CTCAE grade 2 will be excluded as previously indicated.
* Participants who have undergone major systemic surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Participants who are pregnant or breastfeeding.
* Participants with history of known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 12 months of start of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eudocia Q Lee, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - University of California Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - UT, M.D. Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial opened to enrollment on 01/31/17, and the first accrual occurred on 02/09/17. The study permanently closed to accrual on 12/7/22, and the last accrual occurred on 6/18/21. 45 patients were enrolled to the trial with 42 receiving treatment.
Groups:
- Abemaciclib With Surgery (With Postoperative Abemaciclib): * Abemaciclib will be administered on a continuous twice daily dosing schedule
  * Patients who require re-operation will receive a short preoperative course of Abemaciclib
  * Tissue will be used to investigate the ability of Abemaciclib to pass through the blood brain barrier.
  * After recovery from surgery, participants will resume Abemaciclib. Each cycle lasts 28 days.
  * NOTE: enrollment to this arm is complete
  Abemaciclib: Abemaciclib capsule
  Surgery: Surgery
- Abemaciclib Without Surgery: * Abemaciclib will be administered on a continuous twice daily dosing schedule. Each Cycle last 28 days.
  * NOTE: enrollment to this arm is complete
  Abemaciclib: Abemaciclib capsule
- Abemaciclib With Surgery (No Postoperative Abemaciclib): * Abemaciclib will be administered on a continuous twice daily dosing schedule
  * Patients who require re-operation will receive a short preoperative course of Abemaciclib
  * Tissue will be used to investigate the ability of Abemaciclib to pass through the blood brain barrier.
  * After surgery participants will come off study and pursue standard of care treatments at their treating physician's discretion.
  Abemaciclib: Abemaciclib capsule
  Surgery: Surgery
Period: Overall Study
Arm/Group | Abemaciclib With Surgery (With Postoperative Abemaciclib) | Abemaciclib Without Surgery | Abemaciclib With Surgery (No Postoperative Abemaciclib)
Started | 9 | 32 | 1
Completed | 9 | 31 | 1
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Abemaciclib With Surgery (With Postoperative Abemaciclib): Abemaciclib will be administered on a continuous twice daily dosing schedule. Patients who require re-operation will receive a short preoperative course of Abemaciclib.
  Tissue will be used to investigate the ability of Abemaciclib to pass through the blood brain barrier.
  After recovery from surgery, participants will resume Abemaciclib. Each cycle lasts 28 days.
  NOTE: enrollment to this arm is complete Abemaciclib: Abemaciclib capsule Surgery: Surgery
- Abemaciclib Without Surgery: Abemaciclib will be administered on a continuous twice daily dosing. schedule. Each Cycle last 28 days.
  NOTE: enrollment to this arm is complete Abemaciclib: Abemaciclib capsule
- Abemaciclib With Surgery (No Postoperative Abemaciclib): Abemaciclib will be administered on a continuous twice daily dosing schedule. Patients who require re-operation will receive a short preoperative course of Abemaciclib.
  Tissue will be used to investigate the ability of Abemaciclib to pass through the blood brain barrier.
  After surgery participants will come off study and pursue standard of care treatments at their treating physician's discretion.
  Abemaciclib: Abemaciclib capsule Surgery: Surgery
- Total: Total of all reporting groups
Arm/Group | Abemaciclib With Surgery (With Postoperative Abemaciclib) | Abemaciclib Without Surgery | Abemaciclib With Surgery (No Postoperative Abemaciclib) | Total
Number analyzed (Participants) | 9 | 32 | 1 | 42
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [41 to 75] | 60 [41 to 76] | 59 [59 to 59] | 60 [41 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 1 | 20
  Male | 3 | 19 | 0 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 26 | 1 | 35
  Other | 1 | 3 | 0 | 4
  Asian | 0 | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 9 | 32 | 1 | 42

OUTCOME MEASURES:

1. Primary Outcome: Intratumoral Abemaciclib Concentration
Description: Intratumoral abemaciclib concentration defined as the mean tumor-to-plasma ratio in contrast enhancing tissue. Patients were treated with abemaciclib prior to surgery. Tissue and plasma for analysis of this endpoint were obtained at the time of surgery.
Time Frame: Single time point for each participant for collection of tissue and blood at surgery
Population: This analysis included patients who received abemaciclib prior to surgery, regardless of whether they received postoperative abemaciclib (n=9) or no postoperative abemaciclib (n=1) as per protocol. The surgical cohort of the protocol was amended to end study treatment after surgery.
Measure: Mean (Full Range); unit: ng/mL
Groups:
- Abemaciclib With Surgery (With Postoperative Abemaciclib): Experimental: Abemaciclib with Surgery Abemaciclib will be administered on a continuous twice daily dosing schedule
  Patients who require re-operation will receive a short preoperative course of Abemaciclib
  Tissue will be used to investigate the ability of Abemaciclib to pass through the blood brain barrier.
  After recovery from surgery, participants will resume Abemaciclib.
  Each cycle lasts 28 days.
  Abemaciclib: Abemaciclib capsule
- Abemaciclib With Surgery (Without Postoperative Abemaciclib): Participants who require reoperation will be treated with abemaciclib for 10-14 days prior to surgery. Tissue will be used to further investigate the abilities of Abemaciclib. After surgery participants will come off study and pursue standard of care treatments at their treating physician's discretion.
Arm/Group | Abemaciclib With Surgery (With Postoperative Abemaciclib) | Abemaciclib With Surgery (Without Postoperative Abemaciclib)
Number analyzed (Participants) | 9 | 1
ng/mL | 145 [10.6 to 616] | 10.2 [10.2 to 10.2]

2. Primary Outcome: 6-Month Progression Free Survival (PFS6)
Description: The primary endpoint for the nonsurgical cohort was six-month progression free survival (PFS6). Progression is defined by Response Assessment in Neuro-Oncology criteria for high-grade glioma (RANO-HGG) as > 25% increase in sum of the products of perpendicular diameters of enhancing lesions (over best response or baseline if no decrease) on stable or increasing doses of corticosteroids AND/OR one or more of the following: significant increase in T2/FLAIR non-enhancing lesion on stable or increasing doses of corticosteroids steroids compared to baseline scan or best response following initiation of therapy, not due to co-morbid events (radiation therapy, demyelination, ischemic injury, infection, seizures, post-operative changes, or other treatment effects); any new lesion; clear clinical deterioration not attributable to other causes apart from the tumor; or failure to return for evaluation due to death or deteriorating condition.
Time Frame: 6 months
Population: The primary endpoint for the patients treated with abemaciclib in the nonsurgical cohort was PFS6. This Outcome Measure was pre-specified to only assess the "Abemaciclib Without Surgery" Arm/Group.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Groups:
- Abemaciclib Without Surgery: Abemaciclib will be administered on a continuous twice daily dosing schedule. Each Cycle last 28 days.
  NOTE: enrollment to this arm is complete Abemaciclib: Abemaciclib capsule
Arm/Group | Abemaciclib Without Surgery
Number analyzed (Participants) | 31
Percentage of patients | 9.7 [2.5 to 22.9]

3. Secondary Outcome: pRB Expression Level of Tumor Tissue
Description: Expression of levels of phosphorylated retinoblastoma (Rb) to determine if abemaciclib is modulating the intended pathway
Time Frame: 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Time Frame: 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: PK measurements expressed as Area under the plasma concentration versus time curve (AUC) of Abemaciclib [Time Frame C1D1 (pre-treatment), C2D1, C3D1 and C4D1 (each cycle is 28 days)].
Time Frame: 4 months
Reporting Status: Not Posted

6. Secondary Outcome: Peak Plasma Concentration (Cmax)
Description: PK measurements expressed as Peak Plasma Concentration (Cmax) of Abemaciclib [Time Frame C1D1 (pre-treatment), C2D1, C3D1 and C4D1 (each cycle is 28 days)]
Time Frame: 4 months
Reporting Status: Not Posted

7. Secondary Outcome: Radiographic Response Rate
Description: The proportion of participants with measurable disease who experience complete or partial radiographic response determined by the RANO Criteria
Time Frame: 2 years
Reporting Status: Not Posted

8. Secondary Outcome: Median Progression Free Survival
Description: The time from the start of treatment to disease progression or death from any cause
Time Frame: 2 years
Reporting Status: Not Posted

9. Secondary Outcome: Overall Survival
Description: Time from start of study treatment to death from any cause
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) monitored/assessed up to 2 years. AEs are collected from the time of screening through 30 days following end of study treatment and any AEs meeting serious criteria through 90 days following end of study treatment.
Description: An AE is any undesirable sign, symptom or medical condition that develops or worsens in severity after initiating study treatment or any protocol-specified procedure, regardless of attribution. An SAE is any AE at any dose & regardless of causality that: results in death, is life-threatening, requires or prolongs inpatient hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly or birth defect, or is an important medical event.
Groups:
- Abemaciclib With Surgery: Abemaciclib will be administered on a continuous twice daily dosing schedule Patients who require re-operation will receive a short preoperative course of Abemaciclib Tissue will be used to investigate the ability of Abemaciclib to pass through the blood brain barrier.
  After recovery from surgery, participants will resume Abemaciclib. Each cycle lasts 28 days.
  NOTE: enrollment to this arm is complete Abemaciclib: Abemaciclib capsule Surgery: Surgery
- Cohort 1 Surgery Arm: Participants who require reoperation will be treated with abemaciclib for 10-14 days prior to surgery. Tissue will be used to further investigate the abilities of Abemaciclib. After surgery participants will come off study and pursue standard of care treatments at their treating physician's discretion.
  Abemaciclib: Abemaciclib capsule Surgery: Surgery
Arm/Group | Abemaciclib With Surgery | Abemaciclib Without Surgery | Cohort 1 Surgery Arm
All-Cause Mortality (participants affected / at risk) | 9/9 | 31/32 | 1/1
Serious Adverse Events (participants affected / at risk) | 5/9 | 7/32 | 1/1
Other Adverse Events (participants affected / at risk) | 5/9 | 21/32 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abemaciclib With Surgery (N=9) | Abemaciclib Without Surgery (N=32) | Cohort 1 Surgery Arm (N=1)
Decreased Motivation, Abulia (Nervous system disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Femur repair (Surgical and medical procedures) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0
Brain Abscess (Nervous system disorders) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Positive blood cultures with unknown source (Infections and infestations) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Renal calculi (Renal and urinary disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 2 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 — Muscle Weakness R-Leg
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Urinary Urgency (Renal and urinary disorders) | 0 | 2 | 0
Dysphasia (Nervous system disorders) | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
Death NOS (General disorders) | 0 | 2 | 0
Stroke (Nervous system disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abemaciclib With Surgery (N=9) | Abemaciclib Without Surgery (N=32) | Cohort 1 Surgery Arm (N=1)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 3 | 1
Neutrophil count decreased (Investigations) | 2 | 5 | 0
Platelet count decreased (Investigations) | 0 | 2 | 0
White blood cell decreased (Investigations) | 2 | 6 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT02981940/Prot_SAP_000.pdf